CLINICAL TRIAL: NCT02311920
Title: Phase I Study of Ipilimumab, Nivolumab, and the Combination in Patients With Newly Diagnosed Glioblastoma
Brief Title: Ipilimumab and/or Nivolumab in Combination With Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma or Gliosarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02404; NCI-2014-02404 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN002; PNRG-BN002_R05PAPP02; NRG-BN002 (Other: NRG Oncology); NRG-BN002 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2014-12-08; First posted 2014-12-09 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Gliosarcoma; Supratentorial Glioblastoma
MeSH Terms: conditions — Gliosarcoma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (temozolomide and ipilimumab) (Experimental): Within 5 weeks after completion of chemoradiation, patients receive temozolomide PO on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive ipilimumab IV over 90 minutes once every 4 weeks for 4 courses and then beginning 3 months after course 4 once every 3 months for 4 courses in the absence unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Drug: Temozolomide
- Arm II (temozolomide and nivolumab) (Experimental): Within 5 weeks after completion of chemoradiation, patients receive temozolomide PO on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive nivolumab IV over 60 minutes once every 2 weeks for 16 weeks and then once every 2 weeks for 48 weeks in the absence unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Drug: Temozolomide
- Arm III (temozolomide, nivolumab, ipilimumab) (Experimental): Within 5 weeks after completion of chemoradiation, patients receive temozolomide PO on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive ipilimumab IV over 90 minutes once every 4 weeks for 4 courses and nivolumab IV over 60 minutes once every 2 weeks for 64 weeks in the absence unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Drug: Temozolomide

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm I (temozolomide and ipilimumab); Arm III (temozolomide, nivolumab, ipilimumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
  Arms: Arm II (temozolomide and nivolumab); Arm III (temozolomide, nivolumab, ipilimumab)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase I trial studies the safety and best dose of ipilimumab, nivolumab, or both in combination with temozolomide in treating patients with newly diagnosed glioblastoma or gliosarcoma. Monoclonal antibodies, such as ipilimumab and nivolumab, may block tumor growth in different ways by targeting certain cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known which combination is a better treatment for glioblastoma or gliosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum safe dose of single-agent treatment with ipilimumab, nivolumab and the combination when given with temozolomide during maintenance treatment for newly diagnosed glioblastoma.

SECONDARY OBJECTIVES:

I. Collect and record the side effect profiles for single-agent treatment with ipilimumab, nivolumab, and the combination when given with temozolomide during the maintenance phase for newly diagnosed glioblastoma.

II. Perform pilot studies of immune cells within tumor samples, e.g. phenotyping tumor infiltrating lymphocytes (TILs) by interrogating tumor tissues from diagnostic tumor blocks.

III. Report the number of patients alive at 1 and 2 years after the start of single-agent treatment with ipilimumab, nivolumab, and the combination when given with temozolomide during the maintenance phase for newly diagnosed glioblastoma.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Within 5 weeks after completion of chemoradiation, patients receive temozolomide orally (PO) on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive ipilimumab intravenously (IV) over 90 minutes once every 4 weeks for 4 courses and then beginning 3 months after course 4 once every 3 months for 4 courses in the absence unacceptable toxicity.

ARM II: Within 5 weeks after completion of chemoradiation, patients receive temozolomide PO on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive nivolumab IV over 60 minutes once every 2 weeks for 16 weeks and then once every 2 weeks for 48 weeks in the absence unacceptable toxicity.

ARM III: Within 5 weeks after completion of chemoradiation, patients receive temozolomide PO on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive ipilimumab IV over 90 minutes once every 4 weeks for 4 courses and nivolumab IV over 60 minutes once every 2 weeks for 64 weeks in the absence unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 month, and then every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven diagnosis of glioblastoma or gliosarcoma prior to registration by pathology report
* The tumor must be unifocal, confined to the supratentorial compartment and have undergone a gross total or near gross total resection; this will increase the likelihood that the patient will not require corticosteroids or develop pseudoprogression
* The formalin-fixed, paraffin-embedded (FFPE) tumor tissue block must be available to be sent for retrospective central pathology review after registration
* Patients must be registered within 35 days of completion of chemoradiation
* History/physical examination within 7 days prior to registration
* Patients must have undergone an evaluation by magnetic resonance imaging (MRI) within 35 days of completing radiation and must also be within 7 days prior to registration; MRI must NOT demonstrate tumor progression, but patients with imaging changes consistent with pseudo-progression, stable neurologic function and not needing corticosteroid treatment are eligible
* Karnofsky performance status >= 70 within 7 days prior to registration
* Absolute neutrophil count >= 1,500 cells/mm^3
* Platelet count >= 100,000 cells/mm^3
* Hemoglobin (Hgb) > 9 g/dL (can be achieved with transfusion)
* Blood urea nitrogen (BUN) =< 30 mg/dl
* Serum creatinine =< 1.7 mg/dl
* Total bilirubin (except patients with Gilbert's syndrome, who are eligible for the study but exempt from the total bilirubin eligibility criterion) =< 2.0 mg/dl
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN)
* The patient must have completed chemoradiation (all cohorts) within standards of care established by prior Radiation Therapy Oncology Group (RTOG)/Network Radiotherapy Group (NRG) Oncology studies as follows:

  * Radiation therapy

    * Modality: either 3-dimensional (3D) or intensity-modulated radiation therapy (IMRT), or proton therapy is allowed
    * Time to initiation: radiotherapy must be initiated within or equal to 42 days after surgery
    * Target volumes: target volume definition will be based upon postoperative-enhanced MRI; preoperative imaging should be used for correlation and improved identification, as necessary
    * Dose guidelines: the initial target volume will be treated to 46 Gray (Gy) in 23 fractions; after 46 Gy, the cone-down or boost volume will be treated to a total of 60 Gy, with seven additional fractions of 2 Gy each (14 Gy boost dose)
  * Temozolomide during concomitant radiation therapy

    * Temozolomide must have been administered continuously from day 1 of radiotherapy to the last day of radiation (+/- 3 days to take into consideration holidays) at a daily oral dose of 75 mg/m^2 for a maximum of 49 days (except missed doses due to toxicity)
* The patient must not be on a corticosteroid dose greater than physiologic replacement dosing defined as 30 mg of cortisone per day or its equivalent
* The patient must provide study-specific informed consent prior to study entry
* Echocardiogram (ECHO) cardiogram and cardiology consultation required within 7 days prior to registration for patients with a history of congestive heart failure or cardiovascular disease or history of exposure to cardiotoxic agents who are not already excluded

Exclusion Criteria:

* Definitive clinical or radiologic evidence of progressive disease
* Prior placement of Gliadel wafer or local brachytherapy
* Use of an immunotherapy such as a vaccine therapy, dendritic cell vaccine or intracavitary or convectional enhanced delivery of therapy
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Unstable angina within the last 6 months prior to registration
* Transmural myocardial infarction within the last 6 months prior to registration
* Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >= 2 mm using the analysis of an electrocardiogram (EKG) performed within 7 days prior to registration
* New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to registration
* History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months prior to registration
* Serious and inadequately controlled cardiac arrhythmia
* Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Serious or non-healing wound, ulcer, or bone fracture or history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration, with the exception of the craniotomy for tumor resection
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for additional liver function tests and coagulation parameters are not required for entry into this protocol
* Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol
* Active connective tissue disorders, such as lupus or scleroderma, which in the opinion of the treating physician may put the patient at high risk for immunologic toxicity
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome or chronic inflammatory demyelinating polyneuropathy (CIDP), myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded

  * Of note, patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy
* Pregnancy or lactating females; women of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration
* History of severe hypersensitivity reaction to any monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Immune-related dose-limiting toxicities for the single-agent treatment with ipilimumab | Up to 8 weeks
  The frequency and severity of toxicities will be reported.
Immune-related dose-limiting toxicities for the single-agent treatment with nivolumab | Up to 8 weeks
  The frequency and severity of toxicities will be reported.
Immune-related dose-limiting toxicities for the combination of ipilimumab and nivolumab when given with temozolomide | Up to 8 weeks
  The frequency and severity of toxicities will be reported.

SECONDARY OUTCOMES:
Incidence of adverse events, graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 1 month post-treatment
  Will collect and record the side effect profiles for single-agent treatment with ipilimumab, nivolumab, and the combination when given with temozolomide during the maintenance phase for newly diagnosed glioblastoma.
Biomarker analysis of immune cells within tumor samples using standard immunohistochemistry | Up to 1 month post-treatment
  The results of this battery of assays will be used to obtain pilot data and an assessment of feasibility in obtaining reproducible results in preparation for a subsequent randomized, statistically powered comparative clinical trial.
Number of patients who are alive | 1 year after the start of immunotherapy treatment
  The number of patients who are alive at 1 year will be reported.
Number of patients who are alive | 2 years after the start of immunotherapy treatment
  The number of patients who are alive at 2 years will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Gilbert, Principal Investigator — NRG Oncology
Locations (11):
- United States (11):
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Sloan AE, Winter K, Gilbert MR, Aldape K, Choi S, Wen PY, Butowski N, Iwamoto FM, Raval RR, Voloschin AD, Kamiya-Matsuoka C, Won M, Mehta MP. NRG-BN002: Phase I study of ipilimumab, nivolumab, and the combination in patients with newly diagnosed glioblastoma. Neuro Oncol. 2024 Sep 5;26(9):1628-1637. doi: 10.1093/neuonc/noae058. PMID 38874333
- [Derived] Ranjan S, Quezado M, Garren N, Boris L, Siegel C, Lopes Abath Neto O, Theeler BJ, Park DM, Nduom E, Zaghloul KA, Gilbert MR, Wu J. Clinical decision making in the era of immunotherapy for high grade-glioma: report of four cases. BMC Cancer. 2018 Mar 1;18(1):239. doi: 10.1186/s12885-018-4131-1. PMID 29490632